CLINICAL TRIAL: NCT01301911
Title: A Phase I Study of Cipatinib in Patients With HER2 Positive or Uncertain Advanced Breast Cancer
Brief Title: Study of Cipatinib in Patients With HER2 Positive or Uncertain Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XPTN-Ia-1.0
Record Dates: First submitted 2011-01-28; First posted 2011-02-23 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer, Advanced; Cipatinib; phase I; HER2 positive or uncertain advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cipatinib (Experimental): Each subject will receive a single dose of cipatinib on treatment day 1, followed by 4-day observation period, and then will receive cipatinib once daily in cycles consisting of 21 days.
  Interventions: Drug: Cipatinib

INTERVENTIONS:
Drug: Cipatinib — Cipatinib either at 200, 400, 800, 1200, 1400, 1600 or 1800 mg, p.o. once daily

SUMMARY:
Cipatinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. This study is designed to evaluate the safety and tolerability of cipatinib in patients with HER2 positive or uncertain advanced breast cancer:

1. To evaluate the safety and tolerability of cipatinib, and the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT)
2. To determine the pharmacokinetic profile of cipatinib and its metabolites
3. To assess preliminary antitumor activity
4. To determine preliminary regimen for phase II study
5. To determine the relation of expression of HER-1 and HER-2 to the antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 and ≤ 65 years.
* ECOG performance status of 0 to 1.
* Life expectancy of more than 3 months.
* Histologically or cytologic confirmed HER2 positive or uncertain advanced breast cancer that is not curable with available therapies.
* Screening laboratory values within the following parameters:

  * ANC: ≥ 1.5 x 109/L
  * Platelet count: ≥ 100 x 109/L
  * Hemoglobin: ≥ 9.0 g/dL
  * Serum albumin: ≥ 2.5 g/dL
  * Total bilirubin: ≤ 1.5 x upper limit of normal, ULN
  * ALT and AST: ≤ 1.5 x ULN
  * Serum creatinine: ≤ 1.0 x ULN
  * Creatinie clearnce rate: ≥ 50 mL/min
  * Cholesterol≤7.75 mmol/L and triglyceride≤2.5 x ULN
  * LVEF: ≥ 50%
  * QTcF: < 470 ms
* Recovery from all clinically significant AEs related to prior therapies. Duration from the latest therapy is more than 6 weeks for nitroso or mitomycin, or more than 4 weeks for operation, radiotherapy, cytotoxic agents or molecular targeting.
* Ability or willingness to swallow tablets, no dysfunction of gastrointestinal absorption.
* All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test article. For women of child bearing potential, a negative urine or serum pregnancy test result before initiating cipatinib.
* Signed informed consent.

Exclusion Criteria:

* Subjects with third space fluid that can not be controled by drainage or other methods.
* Steroid treatment for more than 50 days, or in need of long-term use of steroids.
* Subjects with uncontrol hypokalemia and hypomagniesemia before study entry.
* Subjects can not interrupt the using of the drugs that may cause QT prolongation during study.
* Subjects with meningioma, or with active central nervous system metastases as indicated by clinical symptoms.
* Subjects with liver metastases which ALT or AST > 1.5 x ULN.
* Treated or treating with EGFR or HER2 TKIs before study entry.
* Receiving any other antitumor therapy.
* Less than 4 weeks from the last clinical trial.
* Pregnant or breastfeeding women.
* Known history of hypersensitivity to cipatinib or any of it components.
* Ongoing infection (determined by investigator).
* Subjects had any heart disease: coronary artery disease, arrhythmia need to treat, heart failure, LVEF < 50%, and any other heart disease that is determined as unfit for this study by investigator, etc.
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study. Examples include, but are not limited to, hypertension, severe diabetes, or thyroid disease.
* Known history of neurological or psychiatric disease, including epilepsy or dementia.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The maximum-tolerated dose (MTD) regimen of cipatinib will be defined as the maximum dose level at which no more than one subject out of six experiences a dose-limiting toxicity (DLT) after completing one treatment cycle. | 3 weeks

SECONDARY OUTCOMES:
Number of participants with adverse events. | 6 weeks
Cipatinib pharmacokinetic parameters may include AUC, Cmax, Tmax, and t1/2. | 3 weeks
Objective response rate (ORR). | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China